CLINICAL TRIAL: NCT02568189
Title: Randomized Controlled Trial of Inferior Vena Cava Ultrasonography in the Management and Disposition of Pediatric Patients Undergoing Evaluation for Sepsis and Dehydration
Brief Title: Utility of Ultrasound Assessment of the Inferior Vena Cava in Patients With Sepsis and Dehydration
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James W Tsung MD MPH, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 15-1599
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Sepsis; Gastroenteritis; Dehydration
Keywords: Sepsis; Gastroenteritis; Dehydration; Ultrasound; Ultrasonography; Inferior Vena Cava
MeSH Terms: conditions — Sepsis; Gastroenteritis; Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sepsis 1 (Experimental): Sepsis patients receiving SonoSite Maxx Series Ultrasound System ultrasound prior to clinical orders including medication and fluid orders being placed by the treating physician
  Interventions: Device: SonoSite Maxx Series Ultrasound System
- Sepsis 2 (Active Comparator): Sepsis patients having SonoSite Maxx Series Ultrasound System ultrasound performed after clinical orders have been placed by the treating physician
  Interventions: Device: SonoSite Maxx Series Ultrasound System
- Gastroenteritis 1 (Experimental): Patients with gastroenteritis receiving SonoSite Maxx Series Ultrasound System ultrasound prior to having orders placed by treating physician
  Interventions: Device: SonoSite Maxx Series Ultrasound System
- Gastroenteritis 2 (Active Comparator): Patients with gastroenteritis having SonoSite Maxx Series Ultrasound System ultrasound after initial clinical orders are placed by treating physician
  Interventions: Device: SonoSite Maxx Series Ultrasound System

INTERVENTIONS:
Device: SonoSite Maxx Series Ultrasound System — Ultrasound imaging is a non-radiating, non invasive modality to assess many areas of the body including vascular fluid status. By placing the probe on the abdomen and looking at the inferior vena cava the clinician can assess a patient's degree of dehydration. We are evaluating the utility of this diagnostic intervention within the clinical management of patients in the pediatric emergency department.

SUMMARY:
Conduct a randomized, controlled trial looking at how the use of ultrasound analyzing the inferior vena cava impacts the management and outcomes of pediatric emergency department patients undergoing evaluation and treatment of sepsis and gastroenteritis associated dehydration.

DETAILED DESCRIPTION:
Ultrasound is a widely accepted and highly useful clinical tool. It carries the additional advantage of being rapid, painless and non-radiating. It has long been used to assess cardiac output and vascular pathologies. More recently emergency and trauma clinicians have been using it to assess hydration status, shock/sepsis states and fluid responsiveness. Using sonography to look at the inferior vena cava gives clinician a rapid view of vascular collapsibility that has been previously demonstrated to correlate with mean arterial pressure (MAP) and central venous pressure (CVP). Previously, Jones et. al. completed an randomized controlled trial (RCT) in adults greater than age 17 evaluating the goal directed utility of early versus delayed inferior vena cava sonography for patients presenting with non traumatic hypotension to the emergency department. This study found improved outcomes and more accuracy in diagnostic etiology in those undergoing immediate IVC imaging. The study conducts a randomized controlled trial of IVC Ultrasonography in pediatric patients 0-21 year of age.

Patients admitted to the Emergency Department and triggering triage STOP SEPSIS ALERT (based on triage vital signs and chief complaint), vomiting requiring zofran or diarrhea with concern for dehydration/hypovolemia, the treating physician believes would benefit from intravenous fluids, will be eligible for inclusion into this study. The "treating physician" refers to one of the Pediatric Emergency Medicine attendings or fellows, listed as co-investigators. Only if and when a patient or parent expresses interest in participating in the study, the attending or fellow caring for the patient will determine if the patient is eligible. If the patient is eligible, and has no criteria that would exclude them from the study, written informed consent will be obtained from the guardian and assent will be obtained in children > 7 years old. The patient will be enrolled in the study and randomized to either the immediate ultrasonography group (Ultrasound (US) of the Inferior Vena Cava (IVC) first before the clinician fully assesses the patient and places rehydration orders) or the control group (US at 15 minutes into the assessment and management of the patient). The goal will be to assess how the use of ultrasound impacts clinical management and outcomes in patients presenting to the pediatric emergency department with sepsis and dehydration.

ELIGIBILITY:
Inclusion Criteria:

* Trigger triage STOP SEPSIS ALERT (based on triage vital signs and chief complaint)
* Present with vomiting requiring Zofran
* Present with diarrhea with concern for dehydration/hypovolemia

Exclusion Criteria:

* Unstable patients with life-threatening injuries who require ongoing resuscitation
* Patient undergoing traumatic resuscitation

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Tsung, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital Department of Emergency Medicine, New York, New York, United States

REFERENCES:
- [Background] Jones AE, Tayal VS, Sullivan DM, Kline JA. Randomized, controlled trial of immediate versus delayed goal-directed ultrasound to identify the cause of nontraumatic hypotension in emergency department patients. Crit Care Med. 2004 Aug;32(8):1703-8. doi: 10.1097/01.ccm.0000133017.34137.82. PMID 15286547
- See also: Article By Jones on goal directed ultrasound — http://www.ncbi.nlm.nih.gov/pubmed/15286547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Halted when Misclassification of Study Outcome Discovered (Different IVC Collapse criteria on IVC Ultrasound)
Pre-assignment Details: 112 participants and enrolled. 6 participants with inferior vena cava not visualized on ultrasound. These participants were not randomized.
Period: Overall Study
Arm/Group | Sepsis 1 | Sepsis 2 | Gastroenteritis 1 | Gastroenteritis 2
Started | 0 | 0 | 52 | 54
Completed | 0 | 0 | 33 | 36
Not Completed | 0 | 0 | 19 | 18
Not completed — Protocol Violation | 0 | 0 | 19 | 18

BASELINE CHARACTERISTICS:
Population: no enrollment for sepsis arms
Groups:
- Total: Total of all reporting groups
Arm/Group | Sepsis 1 | Sepsis 2 | Gastroenteritis 1 | Gastroenteritis 2 | Total
Number analyzed (Participants) | 0 | 0 | 52 | 54 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] |  |  | 6.93 (6.10) | 7.54 (6.31) | 7.2 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 27 | 26 | 53
  Male |  |  | 25 | 28 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Inferior Vena Cava Status [Count of Participants; unit: Participants]
  IVC Collapse |  |  | 39 | 36 | 75
  No IVC Collapse |  |  | 11 | 17 | 28
  Not Visualized |  |  | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Type of Re-hydration
Description: Type of re-hydration: oral vs. intravenous at the time of disposition from the Emergency Department (ED)
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- Gastroenteritis 1 (Immediate): Patients with gastroenteritis receiving SonoSite Maxx Series Ultrasound System ultrasound prior to having orders placed by treating physician
  SonoSite Maxx Series Ultrasound System: Ultrasound imaging is a non-radiating, non invasive modality to assess many areas of the body including vascular fluid status. By placing the probe on the abdomen and looking at the inferior vena cava the clinician can assess a patient's degree of dehydration. We are evaluating the utility of this diagnostic intervention within the clinical management of patients in the pediatric emergency department.
- Gastroenteritis 2 (Delayed): Patients with gastroenteritis having SonoSite Maxx Series Ultrasound System ultrasound after initial clinical orders are placed by treating physician
  SonoSite Maxx Series Ultrasound System: Ultrasound imaging is a non-radiating, non invasive modality to assess many areas of the body including vascular fluid status. By placing the probe on the abdomen and looking at the inferior vena cava the clinician can assess a patient's degree of dehydration. We are evaluating the utility of this diagnostic intervention within the clinical management of patients in the pediatric emergency department.
Arm/Group | Gastroenteritis 1 (Immediate) | Gastroenteritis 2 (Delayed)
Number analyzed (Participants) | 52 | 54
Participants
  Oral Rehydration | 38 | 45
  IV Rehydration | 14 | 9

2. Primary Outcome: Vascular Access Point
Description: For sepsis arm, Secured second vascular access point- type (Interosseous (IO), second Intravenous (IV), central venous (CV) access) within 15 min of physician evaluation
Time Frame: Day 1
Population: Outcome measure for sepsis arms
Arm/Group | Sepsis 1 | Sepsis 2
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Antibiotic Use
Description: For sepsis arm, antibiotic given within 60 min
Time Frame: 60 minutes
Population: Outcome measure for sepsis arms
Arm/Group | Sepsis 1 | Sepsis 2
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Normal Saline Bolus
Description: For sepsis arm, 60 ml/kg Normal Saline bolus administered within 60 minutes
Time Frame: 60 minutes
Population: Outcome measure for sepsis arms
Arm/Group | Sepsis 1 | Sepsis 2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Disposition Status
Description: Pediatric Intensive Care Unit (PICU), Floor, Discharge
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Gastroenteritis 1 (Immediate) | Gastroenteritis 2 (Delayed)
Number analyzed (Participants) | 52 | 54
Participants
  PICU | 0 | 0
  Floor | 3 | 2
  Discharge | 49 | 52

6. Secondary Outcome: Length of ED Stay (From Sepsis Alert to Admission/Discharge Order Entry)
Time Frame: Time between emergency department registration and disposition (admit, transfer or discharge)
Population: No participants enrolled in Sepsis arms
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sepsis 1 | Sepsis 2 | Gastroenteritis 1 | Gastroenteritis 2
Number analyzed (Participants) | 0 | 0 | 52 | 54
minutes |  |  | 200 (121) | 177 (106)

7. Secondary Outcome: Return ED Visit for Same Illness Within 48 Hours
Description: At greater than 48 hours post emergency department disposition
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Gastroenteritis 1 (Immediate) | Gastroenteritis 2 (Delayed)
Number analyzed (Participants) | 52 | 54
Participants | 0 | 0

8. Secondary Outcome: Survival to Hospital Discharge
Description: For sepsis arm, at time of emergency department or hospital discharge
Time Frame: 30 days
Population: Outcome measure for sepsis arms
Arm/Group | Sepsis 1 | Sepsis 2
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: 30 Day Mortality
Description: Assessed any time after 30 days from emergency department registration date.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Gastroenteritis 1 (Immediate) | Gastroenteritis 2 (Delayed)
Number analyzed (Participants) | 52 | 54
Participants | 0 | 0

10. Secondary Outcome: Left Ventricular Function
Description: For sepsis arm, during emergency department visit
Time Frame: Day 1
Population: Outcome measure for sepsis arms
Arm/Group | Sepsis 1 | Sepsis 2
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Source of Sepsis
Description: For sepsis arm, during emergency department or hospital visit
Time Frame: Day 1
Population: Outcome measure for sepsis arms
Arm/Group | Sepsis 1 | Sepsis 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: No participants enrolled in Sepsis arms
Arm/Group | Sepsis 1 | Sepsis 2 | Gastroenteritis 1 | Gastroenteritis 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/52 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/52 | 0/54
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/52 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2015-05-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT02568189/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT02568189/SAP_001.pdf
  • Informed Consent Form (2015-05-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT02568189/ICF_002.pdf